CLINICAL TRIAL: NCT07101835
Title: Extent of Sensory Blockade After External Oblique Intercostal Block for Postoperative Analgesia in Laparoscopic Sleeve Gastrectomy
Brief Title: EOIB for Laparoscopic Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra Turunc, assistant professor, Ondokuz Mayıs University
Other Study IDs: EOIBLSG
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Pain; Regional Anesthesia; Morbid Obesity
Keywords: external oblique intercostal block; acute pain
MeSH Terms: conditions — Acute Pain; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group EOIB: bilateral EOIB (60 ml, %0.25 bupivacaine, totally) + IV morphine patient-controlled analgesia (PCA)
  Interventions: Procedure: Bilateral ultrasound guided external oblique intercostal block (EOIB); Drug: ıv morphine PCA

INTERVENTIONS:
Procedure: Bilateral ultrasound guided external oblique intercostal block (EOIB) — Bilateral ultrasound-guided EOIB (total of 60 ml, %0.25 bupivacaine) will be performed + IV morphine PCA Patients scheduled for LSG will receive a Bilateral ultrasound guided external oblique intercostal block (EOIB) preoperatively, and sensory block status will be evaluated after 30 minutes.
  Other Names: EOIB
Drug: ıv morphine PCA — ıV PCA of 0,5mg/ml morphine (the bolus dose is 20 μg/kg, the lock-in time of 6-10 minutes, the 4-hour limit is adjusted to be 80% of the calculated total amount).
  Other Names: morphine PCA

SUMMARY:
n obese patients, adequate pain relief in the postoperative period is a crucial parameter that affects patient comfort and hospital stay. Improving patient comfort and recovery quality can be achieved by minimizing undesirable effects such as nausea, vomiting, and inadequate analgesia. This study aimed to evaluate the impact of the external oblique intercostal block on postoperative dermatomal distribution, acute pain scores, and opioid consumption during the first 24 hours after laparoscopic sleeve gastrectomy surgery.

DETAILED DESCRIPTION:
In this observational study, patients undergoing laparoscopic sleeve gastrectomy who received either superficial or deep parasternal intercostal plane blocks were evaluated for sensory distribution. Sensory assessment was conducted by a blinded investigator 30 minutes after block administration. Cold sensation testing was performed using small ice tubes applied to the abdominal wall. Sensations were categorized as Normal, Reduced, or No cold.

A successful block was defined as the loss or reduction of cold sensitivity within the expected dermatomal distribution, whereas a normal cold sensation was considered block failure. Assessments began at the midline, including the epigastric region and trocar insertion sites, and progressed laterally toward the anterior axillary line. The extent of sensory coverage was recorded on the skin surface, and marked dermatomal areas were subsequently subjected to digital analysis.

To evaluate block duration, regression of sensory changes was reassessed at 12 and 24 hours postoperatively using the same cold sensation criteria.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years

Exclusion Criteria:

* Patients who did not sign the informed consent form and did not wish to participate in the study
* Patients with a history of opioid use lasting longer than four weeks
* Patients with chronic pain
* Patients with a history of allergy or hypersensitivity to local anesthetics or opioids
* Presence of severe cardiac, hepatic, or renal disease
* Patients with alcohol or drug addiction
* Conditions contraindicating the application of regional anesthesia
* Patients with severe psychiatric disorders such as psychosis or dementia that limit cooperation
* Block failure identified by dermatomal examination after the procedure
* Patients with a STOP-BANG score > 5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing laparoscopic sleeve gastrectomy
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Extent of Sensory Blockade Measured by Cold Sensation Testing Across the Upper Abdominal Wall Following External Oblique Intercostal Block | 30 minutes after the blocks
  Participants will undergo sensory assessment using a standardized cold sensation test at 30 minutes post-block to evaluate the maximum sensory blockade. The data will be recorded as the area of sensory loss (in cm) along the anterior abdominal wall, and the results will be aggregated to report the maximum area of sensory blockade achieved with the external oblique intercostal block. Cold sensation will be categorized as Normal Cold, Reduced Cold, or No Cold Sensation. A successful block is defined as a complete loss or reduction of cold sensitivity.

SECONDARY OUTCOMES:
Cumulative opioid consumption in the first 24 hours after surgery | Postoperative Day 1
  The secondary outcome will be defined as cumulative opioid consumption during the first 12 hours following surgery, calculated in intravenous morphine milligram equivalents (IV-MME). This will include both PCA-administered morphine and rescue intravenous tramadol, in accordance with the standardized ESAIC conversion guidelines. Patients may request opioids using a PCA device when their NRS score is ≥ 4.
Acute pain scores | Postoperative Day 1
  Pain at rest and while coughing will be assessed by numerical rating scale (NRS) scores at 0, 3, 6, 12, 18, and 24 hours after extubation. The NRS is an 11-point numeric scale that ranges from 0 to 10. The NRS is an 11-point scale consisting of integers from 0 to 10: 0 indicates "no pain" and 10 indicates "the worst pain ever possible." One day before the surgery, all patients will be informed about NRS and instructed on how to use a patient-controlled analgesia device.
The number of patients who required rescue analgesia | Postoperative Day 1
  The number of patients requiring rescue analgesics will be recorded over 24 hours.
The incidences of postoperative nausea and vomiting (PONV) | Postoperative Day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18, and 24 hours after extubation. If a score of 3 or more, ondansetron 4 mg IV will be administered and will repeat after 8 hours if required. The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once.
The number of patients with complications | Postoperative 7 days on an average
  The number of patients has any complications -directly related to the block or the drug used in the block- will be recorded
Regression of Sensory Blockade at 12 and 24 Hours Post-Block | Postoperative Day 1
  Block regression will be evaluated at 12 and 24 hours after block administration using cold sensation testing with ice tubes. The cold sensation will be categorized as Normal Cold, Reduced Cold, or No Cold Sensation. Participants who report Normal Cold sensation will be considered to have experienced block regression.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)